CLINICAL TRIAL: NCT04142398
Title: Investigating Human Papillomavirus (HPV) Infection and HPV-Associated Disease in Indian Men Who Have Sex With Men Who Are HIV-Positive
Brief Title: Incidence of HPV Infection and HPV-Associated Disease in Screening Indian Men Who Have Sex With HIV-Positive Men
Status: Withdrawn | Type: Observational
Why Stopped: Closed due to lack of funding.
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AMC-094; NCI-2016-01347 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-094; AMC-094 (Other: AIDS Malignancy Consortium); AMC-094 (Other: CTEP); R21CA167653 (NIH); UM1CA121947 (NIH)
Record Dates: First submitted 2019-08-29; First posted 2019-10-29 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: HIV Infection; Human Papillomavirus Infection; Human Papillomavirus-Related Carcinoma
MeSH Terms: conditions — HIV Infections; Papillomavirus Infections | interventions — Biopsy; Independent Medical Evaluation; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening (health information collection): Participants receive a questionnaire and undergo a targeted physical and anal clinical exam at months 0, 6, and 12. Participants also undergo a penile skin cell and anal swab at months 0, 6, and 12 for cytology, HPV DNA, and CD4+ T-cell count at months 0 and 6 and HIV viral load testing at months 0 and 12. Participants also undergo HRA and penile clinical exam at month 12.
  Interventions: Other: Cytology Specimen Collection Procedure; Procedure: High Resolution Anoscopy with Biopsy; Other: Laboratory Biomarker Analysis; Procedure: Medical Examination; Procedure: Physical Examination; Other: Questionnaire Administration

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo penile skin cell and anal swab collection
  Other Names: Cytologic Sampling
Procedure: High Resolution Anoscopy with Biopsy — Undergo HRA with biopsy
  Other Names: High Resolution Anoscopy-Monitored Biopsy
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Medical Examination — Undergo anal and penile clinical exam
  Other Names: Exam; Examination; Medical Assessment; Medical Exam; Medical Inspection
Procedure: Physical Examination — Undergo targeted physical exam
  Other Names: Assessment; Physical; Physical Assessment; Physical Exam
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research trial studies the incidence of human papilloma virus (HPV) infection and HPV-associated disease in screening Indian men who have sex with human immunodeficiency virus (HIV)-positive men. Gathering health information over time from Indian men who have sex with men (MSM) may help doctors determine how many HIV -positive MSM develop new HPV infections and how many HIV-positive MSM have HPV related disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the prevalence of HPV-associated premalignant lesions in the anus and penis in Indian HIV-seropositive men who have sex with men (MSM).

SECONDARY OBJECTIVES:

I. Describe risk factors for prevalent premalignant lesions in the anus and penis in Indian HIV-seropositive MSM.

II. Describe the prevalence and incidence of penile and anal HPV infection in Indian HIV-seropositive MSM.

OUTLINE:

Participants receive a questionnaire and undergo a targeted physical and anal clinical exam at months 0, 6, and 12. Participants also undergo a penile skin cell and anal swab at months 0, 6, and 12 for cytology, HPV deoxyribonucleic acid (DNA), and CD4+ T-cell count at months 0 and 6 and HIV viral load testing at months 0 and 12. Participants also undergo high-resolution anoscopy (HRA) and penile clinical exam at month 12.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive, as documented by any licensed HIV test according to the Indian National acquired immune deficiency syndrome (AIDS) Control Organization (NACO) guidelines
* Participants report any sex with a man in the past 6 months
* Participants must speak Hindi, Marathi, or English
* Participants should not have any plans to move out of the area in the next 12 months and commit to attending two additional visits one at 6 months and one at 12 months

Exclusion Criteria:

* Active drug or alcohol use or dependence, or other impairment that, in the opinion of the site investigator, would interfere with adherence to study requirements

  * Participants with impairments that, in the opinion of the site investigator, are temporary, will be asked to return another day for enrollment
* Inability to provide informed consent
* History of a sex change operation that would preclude collection of penile or scrotal specimens

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-seropositive MSM in Mumbai, India
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2027-04-30 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HPV-associated high-grade anal intraepithelial neoplasia (HGAIN) | Baseline
  The proportion of men with HPV 6, 11, 16, and/or 18-associated HGAIN will be calculated. HGAIN is determined by biopsy and HPV typing is based on concurrent DNA analysis of anal swabs.
Prevalence of premalignant lesions of the penis | Baseline
  Will be calculated using proportions and exact 95% binomial CI.
Prevalence and incidence of human papillomavirus (HPV) | Up to 12 months
  Will be estimated for specific types, and for all types combined using the life table approach for incidence. Separate estimates will be made for each anatomical site. Risk factors for site-specific incident infection will be evaluated using regression models for survival events observed in discrete time (e.g. pooled logistic regression), incorporating behavioral and biological predictors measured at baseline, and over time at study visits. Risk factors that will be assessed include behavioral and medical history, CD4+ level, and HIV viral load.

SECONDARY OUTCOMES:
The proportion of men with HGAIN at baseline according to presence and absence of HPV infection (types 6, 11, 16, and/or 18). | Baseline
  The proportion of men with HGAIN at baseline according to presence and absence of HPV infection (types 6, 11, 16, and/or 18) will be calculated. HGAIN is determined by biopsy and HPV typing is based on concurrent DNA analysis of anal swabs .
The proportion of men with premalignant lesions of the penis at baseline according to reported number of sex partners in the last 6 months | baseline
  The proportion of men with premalignant lesions of the penis at baseline according to number of sex partners in the last 6 months will be calculated. Premalignant lesions of the penis are determined by colposcopic magnification and HPV typing is based on concurrent DNA analysis of penile swabs.
The proportion of men with HGAIN at baseline according to reported number of sex partners in the last 6 months | baseline
  The proportion of men with HGAIN at baseline according to number of sex partners in the last 6 months will be calculated. HGAIN is determined by biopsy and HPV typing is based on concurrent DNA analysis of anal swabs.
The proportion of men with premalignant lesions of the penis at baseline according CD4+ level. | baseline
  The proportion of men with premalignant lesions of the penis at baseline according to CD4+ level at baseline will be calculated. Premalignant lesions of the penis are determined by colposcopic magnification and HPV typing is based on concurrent DNA analysis of penile swabs .
The proportion of men with HGAIN at baseline according CD4+ level. | baseline
  The proportion of men with HGAIN at baseline according to CD4+ level at baseline will be calculated. HGAIN is determined by biopsy and HPV typing is based on concurrent DNA analysis of anal swabs.
The proportion of men with premalignant lesions of the penis at baseline according to presence and absence of HPV infection (types 6, 11, 16, and/or 18). | Baseline
  The proportion of men with premalignant lesions of the penis at baseline according to presence and absence of HPV infection (types 6, 11, 16, and/or 18) will be calculated. Premalignant lesions of the penis are determined by colposcopic magnification and HPV typing is based on concurrent DNA analysis of penile swabs .

CONTACTS AND LOCATIONS:
Overall Officials: Joel Palefsky, Principal Investigator — AIDS Malignancy Consortium
Locations (3):
- UCSF Medical Center-Parnassus, San Francisco, California, United States
- India (2):
  - Tata Memorial Hospital, Mumbai
  - Udaan Trust, Mumbai